CLINICAL TRIAL: NCT03779126
Title: Efficacy of Combined Low- and High- Frequency Stimulation in Peripheral Muscle Function During Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Wellington Yamaguti, Wellington Pereira dos Santos Yamaguti, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSL 2017-95
Record Dates: First submitted 2018-11-06; First posted 2018-12-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; Electrical stimulation
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: The subjects will be randomised in four groups: 1) low frequency electrical stimulation (LF), 2) high frequency (HF), low and High frequency (LHF), and sham. The subjects will receive electrical stimulation in quadriceps bilaterally for 60 minutes , three times per week, during two months.
Who Masked: Participant, Investigator
Masking Description: The assessments will be conducted for a second investigator to ensure the blinding of first investigator. The subjects will be randomised in four groups (low frequency, high frequency, low and high frequency and sham stimulation) to ensure the blinding of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active comparator (Experimental): Low frequency electrical stimulation for 60 minutes, three times a week during 60 days.
  Interventions: Device: Electrical stimulation
- Other (Experimental): High frequency electrical stimulation for 60 minutes, three times a week during 60 days.
  Interventions: Device: Electrical stimulation
- Experimental group (Experimental): Low and High frequency electrical stimulation for 60 minutes, three times a week during 60 days.
  Interventions: Device: Electrical stimulation
- Placebo (Placebo Comparator): Placebo electrical stimulation for 60 minutes, three times a week during 60 days. In the intervention groups will be used highest intensity tolerated by the individual, and in the sham will be maintained the minimum intensity after beginning of the perception of the electric current
  Interventions: Device: Electrical stimulation

INTERVENTIONS:
Device: Electrical stimulation — 1) Low frequency electrical stimulation (LF) ; High frequency (HF); Low and High frequency (LHF) ; and sham stimulation. Groups will receive bilaterally electrical stimulation, for 60 minutes, three times a week, during two months.
  Other Names: Low frequency electrical stimulation (LF); High frequency (HF); Low and High frequency (LHF); sham stimulation

SUMMARY:
Chronic kidney disease is a systemic disease that affects not only renal function, but also, several organs, bringing social, psychological and physical impact to the patients under this condition. Due to long periods of inactivity during hemodialysis, electrical stimulation becomes a feasible alternative for development physical activity in these patients. Objective: Assess the efficacy of combined low and high frequency electrical stimulation in peripheral muscle function during hemodialysis. Methods: A randomised double-blind clinical trial with chronic kidney disease patient's under hemodialysis, whose will be allocated in four groups: low frequency electrical stimulation (LF) ; high frequency (HF); low and high frequency (LHF); and sham electrical stimulation. The groups will receive quadriceps application bilaterally, for sixty minutes, three times a week, for two months. In the intervention groups will be used highest intensity tolerated by the individual, and in the sham will be maintained the minimum intensity after beginning of the perception of the electric current. The individuals will be evaluated for anthropometry, functional capacity, quality of life and biochemical parameters.

DETAILED DESCRIPTION:
Patients in the present study will be submitted to an evaluation protocol that must be started after the consent of the responsible medical team, and the patient through the Informed Consent Term. On the first day, patients will be evaluated for their personal antecedents, life habits, inflammatory and nutritional status, quality of life, Medical Research Council (MRC) and biochemical markers. On the second day, anthropometry, body composition and functional capacity will be performed. On the third day, the muscular function will be assessed by isokinetic evaluation. After completing the evaluations, patients will be allocated into four groups: low frequency (LF), high frequency (HF), low and high frequency (LHF), and sham.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease
* Classical hemodialysis
* Over 18 years old
* No pace maker
* Without cognitive or motor deficit
* No regular physical activity in the last six months

Exclusion Criteria:

* Abstention for more than two consecutive sessions or four in total
* Inability to perform the tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assess the improvement of muscle mass | Eight weeks
  The muscle mass will be assessed by electric bioimpedance
Assess the improvement of muscle strength | Eight weeks
  The muscle strength will be assessed using isokinetic by peak torque
Assess the improvement of muscle resistance | Eight weeks
  The muscle resistance will be assessed using isokinetic by fatigue index

SECONDARY OUTCOMES:
Assess the improvement of intervention in quality of life | Eight weeks
  The quality of life will be assessed by kidney disease quality of life-short form questionnaire (KDQOL-SF).It is eighty questions about physical aspects, economical and psychological with 80 items. The range could be from 0 to 100. A less score reflect better quality of life.
Correlate peripheral muscle function using medical research council score with nutritional status | Eight weeks
  Peripheral muscle strength will be assessed by medical research council score. It is a score which measure the muscle strength in six plans of movement with range 0 to 60. Higher values represent a better outcome. The findings will be correlated with biomarkers (urea, creatinine, ferritin, lactate and insulin growth factor 1).
Correlate peripheral muscle function using hand grip with nutritional status | Eight weeks
  Peripheral muscle strength will be assessed by hand grip strength. It is a measure the hand grip strength with range 0 to 120 pounds. Higher values represent a better outcome.The findings will be correlated with biomarkers (urea, creatinine, ferritin, lactate and insulin growth factor 1).
Correlate peripheral muscle function with body composition | Eight weeks
  Peripheral muscle function will be assessed by isokinetic dynamometer and body composition will be assessed by bioimpedance (Fresenius)
Correlate peripheral muscle function with functional capacity | Eight weeks
  Peripheral muscle function will be assessed by isokinetic dynamometer and functional capacity will be assessed by six minute step test.
Assess the improvement of intervention in hemodialysis effusion | Eight weeks
  The hemodialysis efficacy will be assessed by Kt/v
Assess the improvement of intervention in functional capacity | Eight weeks
  Functional capacity will be assessed using six minute step test

CONTACTS AND LOCATIONS:
Overall Officials: Wellington PS Yamaguti, Phd, Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Hospitalsiriolibanes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva VG, Amaral C, Monteiro MB, Nascimento DM, Boschetti JR. Effects of inspiratory muscle training in hemodialysis patients. J Bras Nefrol. 2011 Mar;33(1):62-8. English, Portuguese. PMID 21541465
- [Background] Hirai K, Ookawara S, Morishita Y. Sarcopenia and Physical Inactivity in Patients With Chronic Kidney Disease. Nephrourol Mon. 2016 Apr 26;8(3):e37443. doi: 10.5812/numonthly.37443. eCollection 2016 May. PMID 27570755
- [Background] Eidemak I, Haaber AB, Feldt-Rasmussen B, Kanstrup IL, Strandgaard S. Exercise training and the progression of chronic renal failure. Nephron. 1997;75(1):36-40. doi: 10.1159/000189497. PMID 9031268
- [Background] Kopple JD, Wang H, Casaburi R, Fournier M, Lewis MI, Taylor W, Storer TW. Exercise in maintenance hemodialysis patients induces transcriptional changes in genes favoring anabolic muscle. J Am Soc Nephrol. 2007 Nov;18(11):2975-86. doi: 10.1681/ASN.2006070794. Epub 2007 Oct 17. No abstract available. PMID 17942969
- [Background] Koh KP, Fassett RG, Sharman JE, Coombes JS, Williams AD. Effect of intradialytic versus home-based aerobic exercise training on physical function and vascular parameters in hemodialysis patients: a randomized pilot study. Am J Kidney Dis. 2010 Jan;55(1):88-99. doi: 10.1053/j.ajkd.2009.09.025. Epub 2009 Nov 22. PMID 19932545
- [Background] Klassen A, Racasan S, Gherman-Caprioara M, Kurner B, Blaser C, Bahner U, Heidland A. High-tone external muscle stimulation in endstage renal disease: effects on quality of life in patients with peripheral neuropathy. Clin Nephrol. 2013 Jan;79 Suppl 1:S28-33. PMID 23249530
- [Background] Di Iorio B, Torraca S, Gustaferro P, Fazeli G, Heidland A. High-frequency external muscle stimulation in acute kidney injury (AKI): potential shortening of its clinical course. Clin Nephrol. 2013 Jan;79 Suppl 1:S37-45. PMID 23249532
- [Background] Bruggemann AK, Mello CL, Dal Pont T, Hizume Kunzler D, Martins DF, Bobinski F, Pereira Yamaguti W, Paulin E. Effects of Neuromuscular Electrical Stimulation During Hemodialysis on Peripheral Muscle Strength and Exercise Capacity: A Randomized Clinical Trial. Arch Phys Med Rehabil. 2017 May;98(5):822-831.e1. doi: 10.1016/j.apmr.2016.12.009. Epub 2017 Jan 16. PMID 28093194
- [Background] Sesso RC, Lopes AA, Thome FS, Lugon JR, Martins CT. Brazilian Chronic Dialysis Census 2014. J Bras Nefrol. 2016 Mar;38(1):54-61. doi: 10.5935/0101-2800.20160009. English, Portuguese. PMID 27049365
- [Background] Hays RD, Kallich JD, Mapes DL, Coons SJ, Carter WB. Development of the kidney disease quality of life (KDQOL) instrument. Qual Life Res. 1994 Oct;3(5):329-38. doi: 10.1007/BF00451725. PMID 7841967
- [Background] Duarte PS, Ciconelli RM, Sesso R. Cultural adaptation and validation of the "Kidney Disease and Quality of Life--Short Form (KDQOL-SF 1.3)" in Brazil. Braz J Med Biol Res. 2005 Feb;38(2):261-70. doi: 10.1590/s0100-879x2005000200015. Epub 2005 Feb 15. PMID 15785838
- [Background] Franssen FM, Broekhuizen R, Janssen PP, Wouters EF, Schols AM. Limb muscle dysfunction in COPD: effects of muscle wasting and exercise training. Med Sci Sports Exerc. 2005 Jan;37(1):2-9. doi: 10.1249/01.mss.0000150082.59155.4f. PMID 15632660
- [Background] Hough CL, Lieu BK, Caldwell ES. Manual muscle strength testing of critically ill patients: feasibility and interobserver agreement. Crit Care. 2011;15(1):R43. doi: 10.1186/cc10005. Epub 2011 Jan 28. PMID 21276225
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E. Normative data for grip strength of elderly men and women. Am J Occup Ther. 1995 Jul-Aug;49(7):637-44. doi: 10.5014/ajot.49.7.637. PMID 7573334
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] Breitsameter G, Figueiredo AE, Kochhann DS. Calculation of Kt/V in haemodialysis: a comparison between the formulas. J Bras Nefrol. 2012 Mar;34(1):22-6. English, Portuguese. PMID 22441178
- [Background] Keane D, Gardiner C, Lindley E, Lines S, Woodrow G, Wright M. Changes in Body Composition in the Two Years after Initiation of Haemodialysis: A Retrospective Cohort Study. Nutrients. 2016 Nov 4;8(11):702. doi: 10.3390/nu8110702. PMID 27827911
- [Background] Arcuri JF, Borghi-Silva A, Labadessa IG, Sentanin AC, Candolo C, Pires Di Lorenzo VA. Validity and Reliability of the 6-Minute Step Test in Healthy Individuals: A Cross-sectional Study. Clin J Sport Med. 2016 Jan;26(1):69-75. doi: 10.1097/JSM.0000000000000190. PMID 25706661
- [Background] Pessoa BV, Arcuri JF, Labadessa IG, Costa JN, Sentanin AC, Di Lorenzo VA. Validity of the six-minute step test of free cadence in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2014 May-Jun;18(3):228-36. doi: 10.1590/bjpt-rbf.2014.0041. PMID 25003275
- [Background] Segers J, Hermans G, Bruyninckx F, Meyfroidt G, Langer D, Gosselink R. Feasibility of neuromuscular electrical stimulation in critically ill patients. J Crit Care. 2014 Dec;29(6):1082-8. doi: 10.1016/j.jcrc.2014.06.024. Epub 2014 Jun 30. PMID 25108833
- [Background] Parry SM, Berney S, Warrillow S, El-Ansary D, Bryant AL, Hart N, Puthucheary Z, Koopman R, Denehy L. Functional electrical stimulation with cycling in the critically ill: a pilot case-matched control study. J Crit Care. 2014 Aug;29(4):695.e1-7. doi: 10.1016/j.jcrc.2014.03.017. Epub 2014 Mar 26. PMID 24768534
- [Result] Dobsak P, Homolka P, Svojanovsky J, Reichertova A, Soucek M, Novakova M, Dusek L, Vasku J, Eicher JC, Siegelova J. Intra-dialytic electrostimulation of leg extensors may improve exercise tolerance and quality of life in hemodialyzed patients. Artif Organs. 2012 Jan;36(1):71-8. doi: 10.1111/j.1525-1594.2011.01302.x. Epub 2011 Aug 16. PMID 21848929
- [Derived] de Souza Francisco D, Moraes IG, Brito CP, Righetti RF, Yamaguti WP. The phase angle cut-off point capable of discriminating hemodialysis patients with reduced exercise tolerance: a cross-sectional study. BMC Sports Sci Med Rehabil. 2024 Feb 2;16(1):34. doi: 10.1186/s13102-024-00825-5. PMID 38308310
- [Derived] Moraes IG, Brito CP, Francisco DS, Faria LM, Luders C, de Brito CMM, Yamaguti WP. Efficacy of neuromuscular electrical stimulation with combined low and high frequencies on body composition, peripheral muscle function and exercise tolerance in patients with chronic kidney disease undergoing haemodialysis: a protocol for a randomised, double-blind clinical trial. BMJ Open. 2022 Nov 9;12(11):e062062. doi: 10.1136/bmjopen-2022-062062. PMID 36351736